CLINICAL TRIAL: NCT07362927
Title: An Exploratory Clinical Study Evaluating LX111 Gene Therapy in Patients With Diabetic Macular Edema (DME)
Brief Title: Safety and Efficacy Evaluation of LX111 Gene Therapy in DME Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LX111-01
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Macular Edema (DME)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LX111 Dose Escalation up to 2 dose levels (Experimental): Qualified participants will receive a single unilateral intravitreal injection of LX111 at Day 0.
  Interventions: Genetic: LX111 Injection
- LX111 Dose Expansion Dose 1 (Experimental): Qualified participants will receive a single unilateral intravitreal injection of LX111 at Day 0.
  Interventions: Genetic: LX111 Injection
- LX111 Dose Expansion Dose 2 (Experimental): Qualified participants will receive a single unilateral intravitreal injection of LX111 at Day 0.
  Interventions: Genetic: LX111 Injection

INTERVENTIONS:
Genetic: LX111 Injection — LX111 is an rAAV gene therapy vector carrying a coding sequence for VEGF-trap.

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of LX111 treatment of DME. This study will enroll participants aged ≥ 18 vears old to receive a single unilateral intravitreal (lVT) injection of LX111 to evaluate its safety and efficacy.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, dose-ranging trial to evaluate the safety and efficacy of LX111 in participants with DME. The trial will be conducted in two parts: Dose Confirmation and Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent, and willing to attend follow-up visits;
2. Age ≥ 18;
3. Type I or Type II diabetes mellitus with macular thickening secondary to DME involving the center of the fovea;
4. CST ≥ 300 μm in the study eye at Screening;
5. BCVA ETDRS letters between 19 and 73;
6. Participants must have received anti-VEGF therapy within 12 months prior to screening and demonstrated a meaningful response;
7. Male subjects whose partner is a fertile female or female subjects who are fertile, agree to take effective contraceptive measures from the screening period until the last follow-up.

Exclusion Criteria:

1. Active proliferative diabetic retinopathy (PDR);
2. Presence of iris neovascularization in the study eye at Screening;
3. Retinal laser photocoagulation in the study eye within 3 months prior to Screening;
4. Prior gene therapy in the study eye;
5. The study eye has been treated with an intravitreal dexamethasone implant (Ozurdex®) within 6 months prior to Screening.
6. Systemic anti-VEGF treatment within 3 months before Screening;
7. Received an investigational drug, agent, device, or therapy (ocular or non-ocular) in the 3 months (or at least 5 half-lives, whichever is longer) prior to Screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events in the eyes and throughout the body within 364 days after LX111 treatment | 52 weeks
  Incidence of adverse events and serious adverse events within 52 weeks of LX111 intravitreal injection in each dose group.
Dose Limiting Toxicity | 4 weeks
  The incidence of DLT in each dose group.

SECONDARY OUTCOMES:
Mean changes in BCVA from Baseline | 12 weeks, 36 weeks, 52 weeks
  The mean changes of BCVA scores on the ETDRS chart at different timepoints after LX111 treatment compared with baseline.
Mean changes in Central Subfield Thickness (CST) from Baseline | 12 weeks, 36 weeks, 52 weeks
  The mean changes of CST at different timepoints after LX111 treatment compared with baseline.
The percentage of participants who received anti-VEGF supplemental injection within 52 weeks after LX111 treatment | 52 weeks
  The proportion of participants who received anti-VEGF supplemental injection within 52 weeks after LX111 treatment
Proportion of participants achieving an improvement or worsening in DR in the study eye per the ETDRS-DRSS on ultra-wide field fundus photography. | 52 weeks
  To evaluate the effect of LX111 on DR (ETDRS-DRSS) over time.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai
  - Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No